CLINICAL TRIAL: NCT04314011
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Study of Umbilical Cord Mesenchymal Stem Cells Infusion for Aging Frailty
Brief Title: Clinical Study of Umbilical Cord Mesenchymal Stem Cells Infusion for Aging Frailty
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EC.D (BG).020.02.0
Record Dates: First submitted 2019-12-10; First posted 2020-03-18 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Aging Frailty

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HUC-MSCs Group (Experimental): Human umbilical cord mesenchymal stem cells (1*10^6/kg cells): delivered via peripheral intravenous infusion.
  Interventions: Biological: Human umbilical cord mesenchymal stem cells（HUC-MSCs）
- Control Group (Placebo Comparator): Placebo:normal saline delivered via peripheral intravenous infusion.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Human umbilical cord mesenchymal stem cells（HUC-MSCs） — Human umbilical cord mesenchymal stem cells（HUC-MSCs）
  Arms: HUC-MSCs Group
Biological: Placebo — Placebo
  Arms: Control Group

SUMMARY:
The purpose of this clinical study is to answer the questions:

1. Is the proposed intervention safe?
2. Is the proposed intervention effective in improving the healthy status of subjects with aging frailty?

DETAILED DESCRIPTION:
Aging frailty is a clinical syndrome, characterized by a decrease of homeostatic reserves and enhanced vulnerability to endogenous or exogenous stressors, exposing individuals to an increased risk of adverse health-related outcomes. The human umbilical cord (HUC) is a promising source of mesenchymal stem cells (MSCs), compared to embryonic stem cells, HUC-MSCs are noncontroversial with a painless collection procedure and faster self-renewal properties. HUC-MSCs can differentiate into the different germ layers and modulate immune responses. One possible mechanism for the onset and development of aging frailty is the depletion of stem cells. Hence, intravenous infusion of HUC-MSCs is attractive therapy against aging frailty.

This is a randomized, double-blind, placebo-controlled clinical trial. The participants (n = 30) will be randomly distributed into two groups. The HUC-MSCs Group (n = 15) will receive intravenous infusion of mesenchymal stem cells twice over a month (30 days interval), the Control Group (n = 15) will receive the same protocolized intervention with normal saline. Follow-up duration is 6 months after first intervention. The reported serious adverse events（SAEs）will be observed within one month post infusion. The short-item from health survey（SF-36), EuroQol five dimensions questionnaire (EQ-5D) and Fried phenotype scale will be evaluated. Short physical performance battery (SPPB) and plasm biomarkers will be assessed.The assessments will be performed at baseline, 1 month, 3 months and 6 months.

The intent of this study is to explore domains of efficacy of HUC-MSCs through the reduction of signs and symptoms of aging frailty and to evaluate the safety of HUC-MSCs in subjects with aging frailty.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age ≥60 and ≤80 years at the time of signing the informed consent form.
2. Must show signs of frailty apart from a concomitant condition as assessed by the investigator with a frailty score of 1 to 4 using the Fried Phenotype Scale.
3. Must provide written informed consent.
4. Subjects are expected to live more than 12 months.

Exclusion Criteria:

1. Serious comorbid illness that, in the opinion of the investigator, may compromise the safety or compliance of the patient or preclude successful completion of the study
2. Advanced liver or renal failure, class III/IV congestive heart failure, myocardial infarction, unstable angina, cardiac revascularization, or severe obstructive ventilator defect.
3. Uncontrolled hypertension or hyperglycemia.
4. Have known allergies to biological drugs or antibiotics.
5. Expecting to receive organ transplantation.
6. Have a clinical history of malignancy or active autoimmune diseases.
7. Have a history of drug or alcohol abuse within the past 24 months.
8. Be serum-positive for HIV, hepatitis BsAg or viremic hepatitis C.
9. Be currently participating (or participated within the previous 30 days) in an investigational therapeutic or device trial.
10. Be a female who is pregnant, nursing, or of childbearing potential while not practicing effective contraceptive methods.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Safety of HUC-MSCs infusion | Within one month post infusion
  Safety were assessed by incidence of reported serious adverse events (SAEs) within one month after infusion. An SAE is defined as any untoward medical occurrence that:
  1. Results in death
  2. Is life-threatening (stroke or non-fatal pulmonary embolism, etc.)
  3. Requires inpatients hospitalization or prolongation of hospitalization
  4. Results in clinically significant abnormal laboratory test results or abnormal vital signs, based on clinical judgment.

SECONDARY OUTCOMES:
Difference in rate of decline of Frailty | Baseline, month 1, 3 month and 6 months post infusion
  Difference in rate of decline of Frailty assessed using Fried phenotype scale:
  1. Slowing of Mobility (assessed via a 4-meter gait speed test; Timed up and go (TUG) test and Short Physical Performance Battery (SPPB) assessment)
  2. Weight Loss (assessed via weighing scale)
  3. Reduced Activity (assessed via Minnesota Leisure Time Activities (MLTA) questionnaire)
  4. Diminished handgrip strength (assessed via dynamometer)
  5. Exhaustion (assessed by two items from the Center for Epidemiological Studies-Depression, CES-D):" I felt that everything I did was an effort? and I could not get going."
Difference in subject quality of life assessments | Baseline, month 1, month 3 and month 6 post infusion
  Health-related quality of life will be assessed via Short-Form 36 Health Survey (SF-36), including physical functioning scale and mental health index; the health status including Health State Index (HSI) and respondent's self-rated health on a vertical scale will be accessed via EuroQol 5-Dimension (ED-5D).
Changes in the pro-inflammatory cytokines of blood sample between the HUC-MSC and placebo cohorts | Baseline, month 1, month 3 and month 6 post infusion
  Enzyme-linked immunosorbent assay will be used to identify the serum levels of pro-inflammatory cytokines (e.g.,Interleukin-6).
Changes in cellular components of the immune system between the HUC-MSC and placebo cohorts | Baseline, month 1, month 3 and month 6 post infusion
  Flow cytometry will be used to identify the changes in numbers of lymphocyte subpopulations (e.g., B cells, T cells).

CONTACTS AND LOCATIONS:
Overall Officials: Zhongming Liu, MD/Ph.D, Principal Investigator — Shanghai East Hospital, Shanghai Tongji University
Locations (1):
- Shanghai East Hospital, Shanghai Tongji University, Shanghai, China

REFERENCES:
- [Derived] Zhu Y, Huang C, Zheng L, Li Q, Ge J, Geng S, Zhai M, Chen X, Yuan H, Li Y, Jia W, Sun K, Li Y, Ye T, Zhao Z, Liu H, Liu Z, Jiang H. Safety and efficacy of umbilical cord tissue-derived mesenchymal stem cells in the treatment of patients with aging frailty: a phase I/II randomized, double-blind, placebo-controlled study. Stem Cell Res Ther. 2024 Apr 29;15(1):122. doi: 10.1186/s13287-024-03707-2. PMID 38679727